CLINICAL TRIAL: NCT03032991
Title: Early Biomarkers of Neurodevelopment in Offspring of Diabetic Mothers (GD-BRAIN)
Brief Title: Early Biomarkers of Neurodevelopment in Offspring of Diabetic Mothers
Acronym: GD-BRAIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Murcia (Other)
Collaborators: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Elvira Larqué, Professor, Universidad de Murcia
Other Study IDs: SAF2015-69265
Record Dates: First submitted 2017-01-13; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Gestational Diabetes Mellitus in Childbirth; Neurodevelopmental Disorders
Keywords: Gestational diabetes; Neurodevelopment; Placenta; Gut microbiota; Protectins; MFSD2a; AdipoRon
MeSH Terms: conditions — Neurodevelopmental Disorders; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Children at 8 years old born from healthy pregnancies
- GDM: Children at 8 years old born from mothers with gestational diabetes during pregnancy

SUMMARY:
The prospective multicenter study GD-Brain provides a better knowledge on the basis of neurological impairment in children born to mothers with gestational diabetes (GDM). GDM modifies placental structure and affect materno-fetal nutrient transfer. Docosahexaenoic acid (DHA) play an important role on neurodevelopment, and it is reduced in venous cord blood of newborns born to GDM. In previous studies, we have already demonstrated impaired DHA fetal levels not only using label fatty acids with stable isotopes administrated to pregnant women, but also in observational studies in GDM as the prevention of obesity study (PREOBE study) in Granada and other similar study in Murcia. The impaired cord DHA levels were associated to disturbed neurodevelopment in these children during the first year of life. However, it is uncertain the mechanisms underlying this impaired materno-fetal DHA transfer and implications for later life.

The recent publication in Nature Journal of a selective transmembrane carrier for DHA in brain named "major facilitator superfamily domain 2a" (MFSD2a) open new expectations. We detected disturbed MFSD2a levels in placentas from GDM which could be due to structural problems in this organ; inflammation, oxidation and metabolic changes related to diabetes might affect MFSD2a activity. Moreover, it is difficult to know whether disturbed MFSD2a levels in placenta may also indicate altered levels of this carrier in the brain from children born to GDM mothers, which could contribute to neurodevelopment impairment in these subjects. Recent studies also indicate that obesity alters the biosynthesis of eicosanoids derived from DHA, with a decrease of protectins and resolvin of D-series, which have powerful anti-inflammatory properties.

The main aim of this study is to analyse potential differences on neurodevelopment, and brain structure and functioning, in children 8 years old born to GDM respect to those born to healthy normoweight mothers, as well as to identify early biomarkers consistently related to neurodevelopment from early stages of life.

DETAILED DESCRIPTION:
We will contact to participants from the PREOBE study and Murcia's cohorts study to get involved a total of 174 children at 8 years of age. The results from neurodevelopment evaluation by neuropsychological testing, neurological functions rhythms and neuroimaging (fMRI and DTI) at 8 years old will be associated to clinical and metabolic data recorded during pregnancy.

As secondary aim, we would discern whether the decrease on DHA levels in offspring of GDM at birth is associated to disturbed neurodevelopment at 8 years old.

The impact of maternal diabetes on placental MFSD2a and children's resolvin and protectins derived from DHA will be measured in urine samples at 8 years old.

Gut microbiota composition and function will be also studied to detect its role in the potential disturbances regarding the production of anti-inflammatory mediators.

A part from the clinical study, we will perform an intervention trial using animal models. Gestational rats with diabetes and control rats will be treated with antioxidants and adipoRon in order to delay neuro-degeneration in these animals because of the diabetes, as well as their influence on MFSD2a levels in placenta and brain. All these studies may provide to the industry of valuable information to improve nutritional supplements during gestation or infancy to avoid potential delay of cognitive functions in offspring of diabetic mothers.

ELIGIBILITY:
Inclusion Criteria:

* Children from healthy pregnancies and GDM pregnancies from the ^PREOBE study and GDM Murcia study.

Exclusion Criteria:

-

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 174 Children born between 2008-2011 from 2 previous studies:
  * PREOBE study from the University of Granada
  * GDM Murcia study from the University of Murcia
Sampling Method: Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological battery | 8 years old
  Neuropsychological battery to cover different neuropsychological domains: processing speed, memory, attention, language, executive functions, and behaviour (parent-completed measure).
Neuroimaging ( functional MRI) | 8 years
  Anatomical magnetic resonance imaging (fMRI)
Electroencephalography (EEG) | 8 years
  Stereotyped electrophysiological response to several external stimulus

SECONDARY OUTCOMES:
Fatty acids | 8 years old
  Fatty acid profile in oral mucose
Metabolomic | 8 years old
  Prostaglandins, thromboxans, isoprostanes, resolvin in urine samples

OTHER OUTCOMES:
Microbiome | 8 years old
  Metagenome
Maturation of circadian rhythm | 8 years old
  Analysis of the circadian rhythm of temperature, activity and sleep
Nutritional evaluation | 8 years old
  Dietary assessment by food frequency questionnaire and by 3 day of dietary record
Physical activity | 8 years old
  questionnaires
Physical Activity | 8 years old
  Accelerometers will be used also to record activity of the subjects

CONTACTS AND LOCATIONS:
Overall Officials: Elvira Larqué, Dr., Principal Investigator — Universidad de Murcia; Cristina Campoy, MD, Principal Investigator — Universidad de Granada
Locations (1):
- Elvira Larqué, Murcia, Murcia, Spain